CLINICAL TRIAL: NCT03648476
Title: Intervention to Change Attributions That Are Negative (ICAN): a New Approach to Reducing Anger and Aggression After Brain Injury
Brief Title: Intervention to Change Attributions That Are Negative (ICAN)
Acronym: ICAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dawn Neumann, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1806829789; 1R21HD094232-01 (NIH)
Record Dates: First submitted 2018-08-20; First posted 2018-08-27 (Actual); Results first posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Trauma, Brain; Brain Injuries; Traumatic Brain Injury; Brain Injuries, Traumatic; Brain, Trauma
Keywords: Anger; Aggression; Hostility
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Aggression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICAN (Experimental): 6-week group therapy intervention with clinical RA comprised of 6 90-120 minute sessions beginning after Time 1 testing
  Interventions: Behavioral: ICAN
- WLC: Waitlist Control (Other): WLC participants will delay treatment until after time two testing 8-weeks from time one testing. Participants will then begin 6 90-120 minute therapy sessions.
  Interventions: Behavioral: ICAN

INTERVENTIONS:
Behavioral: ICAN — A 6-week group therapy sessions once a week for 90-120 minutes.

SUMMARY:
ICAN is the first treatment to target hostile attributions after TBI, making it a novel anger/ aggression management approach in this population. This is a randomized waitlist control trial. The length of time in the trial is approximately 15 weeks and the intervention is 6 weeks long.

DETAILED DESCRIPTION:
ICAN is the first treatment to target hostile attributions after TBI, making it a novel anger/ aggression management approach in this population. Since the investigator's prior research shows that stronger hostile attributions are associated with poorer perspective taking,39 ICAN employs a unique perspective-positioning technique to train perspective taking and reduce hostile attributions. After recalling a personal situation in which others' ambiguous actions led to an unpleasant outcome, participants will explore different perspectives: sitting or standing in one position, s/he will explore his or her own thoughts and feelings (self-perspective), then move to a different position to experience the other person's perspective, eliciting their thoughts and feelings.

In 40 participants with TBI, we will conduct a Phase I, randomized waitlist controlled trial with 4 data collection points: Baseline; Week 1; Week 8 (post-treatment for ICAN; post-wait period for WLC); Week 15 (WLC post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* History of complicated mild to severe TBI (injury due to an external physical force), with injury severity being defined either by Glasgow Coma Score at time of injury (≤12), or post-traumatic amnesia (≥1 day), or loss of consciousness (≥30 minutes), or positive head CT scan consistent with TBI.
* At least 18 years of age or older;
* ≥1 year post-injury;
* Have adequate vision, hearing, and speech/ language skills to participate in assessments and group therapy (determined based on interaction with the participant at screening)
* Have adequate reading comprehension (due to the primary assessment involving written scenarios)
* Have abnormal scores of negative attributions or perspective taking (determined at T0 screening)
* Have above average aggression (prescreened on telephone, and confirmed T0 screening).
* No anticipated medication changes for emotions/ behavior during length of study participation; medications for emotions/ behavior must be stable within last 30 days prior to consent at T0 (Screening)
* Have reliable mode of transportation

Exclusion criteria:

* Pre-morbid neurological disorders that could affect mood and cognition (e.g. stroke); does not include controlled seizures
* Progressive central nervous system disorders (e.g. dementia, Parkinson's)
* Developmental disability (e.g., autism, developmental delay);
* Major psychiatric disorders (e.g. schizophrenia, Borderline Personality Disorder);
* Severe Depression and/or perceived risk to self or others (mental health resources will be provided and if suicide risk, approved suicide protocol will be utilized);
* Currently receiving active behavioral therapy for anger.
* On drug research study for irritability, anger, aggression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Neumann, Phd, Principal Investigator — Indiana University School of Medicine
Locations (1):
- The Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants were enrolled (signed consent); however, 4 participants withdrew from the study PRIOR to randomization to the study arm.
Period: Overall Study
Arm/Group | ICAN | WLC: Waitlist Control
Started | 10 | 14
Completed | 8 | 13
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICAN | WLC: Waitlist Control | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.7) | 43.1 (12.7) | 42 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Buss-Perry Aggression Questionnaire Score
Description: The Buss-Perry Aggression Questionnaire (AQ), is a standardized measure comprised of 34 statements to assess total aggression, as well as the following aggression subconstructs: anger, hostile thoughts, and physical and verbal aggression. Participants rate statements using a 5-point Likert scale (1, 2, 3, 4, 5).
  Subscales are summed to compute a Total Aggression raw score and total Aggressions Scores were then converted to T scores (1-100) with a mean T-score =50 and Standard deviation=10 points.
  Higher T-scores= more aggression/ worse outcome, thus a lower number indicates improvement Here, we are reporting the CHANGE in the group's MEAN t-score (e.g. Mean Post-test T score of 62 MINUS Mean Pre-test t score of 58 = Mean CHANGE score of -4, which means less aggression post-treatment). Thus, we are NOT reporting t-scores in this Results section; just the mean change of these scores. Negative scores indicate an improvement.
Time Frame: Change from Baseline at Week 8 and Week 15
Population: Week 8 is post-intervention for ICAN, where as WLC had not yet received the intervention. Only WLC subjects were tested at Week 15, and that is their post-test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ICAN | WLC: Waitlist Control
Number analyzed (Participants) | 8 | 13
score on a scale
  Change from Baseline to Week 8 | -1.7 (.27) | -5.91 (3.6)
  Change from baseline to week 15: number analyzed (Participants) | 0 | 13
  Change from baseline to week 15 |  | -8.51 (1.32)

2. Secondary Outcome: Change in Anger Affect Score
Description: The Anger-Affect Scale, from the PROMIS Anger, is a 5 item subjective questionnaire that requires participants to indicate the frequency with which they have been bothered by anger symptoms in the past week using a 5 point Likert scale (1.2,3,4,5). Total Raw scores range from 5-25. Higher scores indicate more severe anger; lower scores indicate lower levels of anger. Thus, a negative change score indicates a reduction in anger.
Time Frame: Change from Week 1 at Week 8 and Week 15
Population: Week 8 is post intervention for ICAN, but WLC will not have received the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ICAN | WLC: Waitlist Control
Number analyzed (Participants) | 8 | 13
score on a scale
  Change from Baseline to Week 8 | -1.95 (.19) | -.89 (2.17)
  Change from Baseline to Week 15: number analyzed (Participants) | 0 | 13
  Change from Baseline to Week 15 |  | -4.49 (1.63)

3. Secondary Outcome: Global Impression of Change for Anger and Aggression
Description: The Global Impression of change for Anger and Aggression is a 1 item question that measures perceived change in anger and aggression Using a 7-point scale (1="no change" to "A great deal better, and a considerable improvement that has made all the difference"). Total Raw scores range from 1-7.Higher scores indicate greater change.
  1. No change (or condition has gotten worse)
  2. Almost the same, hardly any change at all
  3. A little better, but no noticeable change
  4. Somewhat better, but the change has not made any real difference
  5. Moderately better, and a slight but noticeable change
  6. Better, and a definite improvement that has made a real and worthwhile difference
  7. A great deal better, and a considerable improvement that has made all the difference
Time Frame: Week 8 for participants randomized to ICAN or Week 15 for those randomized to WLC (administered after receiving treatment)
Population: This assessment was sent to the participants electronically. There is missing data from one participant who was randomized to ICAN. All participants (ICAN and WLC) had received the intervention by the time this outcome assessment was administered.
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- WLC (Post-intervention): WLC participants will delay treatment until after time two testing 8-weeks from time one testing. Participants will then begin 6 90-120 minute therapy sessions.
  After wait period, participants in the WLC receive the ICAN treatment.
  ICAN: A 6-week group therapy sessions once a week for 90-120 minutes.
Arm/Group | ICAN | WLC (Post-intervention)
Number analyzed (Participants) | 7 | 13
score on a scale | 4 (1.90) | 4 (1.98)

4. Secondary Outcome: Global Impression of Change for Perspective Taking and Empathy
Description: The Global Impression of change for Perspective Taking and Empathy is a 1 item question that measures perceived change in Perspective Taking and Empathy using a 7-point scale (1="no change" to "A great deal better, and a considerable improvement that has made all the difference"). Total Raw scores range from 1-7.Higher scores indicate greater change.
  1. No change (or condition has gotten worse)
  2. Almost the same, hardly any change at all
  3. A little better, but no noticeable change
  4. Somewhat better, but the change has not made any real difference
  5. Moderately better, and a slight but noticeable change
  6. Better, and a definite improvement that has made a real and worthwhile difference
  7. A great deal better, and a considerable improvement that has made all the difference
Time Frame: Week 8 for participants randomized to ICAN or Week 15 for those randomized to WLC (administered after received treatment)
Population: This assessment was sent to the participants electronically. There is missing data from several participants who did not return their survey after multiple attempts (ICAN missing data=1; WLC missing data=8). All participants (ICAN and WLC) had received the intervention by the time this outcome assessment was administered.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | ICAN | WLC (Post-intervention)
Number analyzed (Participants) | 7 | 5
score on a scale | 5 (1.15) | 6 (.55)

5. Other Pre Specified Outcome: Change in Interpersonal Reactivity Index (IRI) - Perspective Taking and Empathic Concern Score
Description: We will use 2 subscales from the Interpersonal Reactivity Index: Perspective-taking and Empathic Concern. It is a standardized, subjective measure that uses a 5 point scale. There are 7 questions for each subscale.
  Scale (0,1,2,3,4). Scores are calculated each subscale Perspective scale scores range from 0-28 Empathic concern scores range from 0-28 Higher scores indicate more perspective taking and empathy
Time Frame: Change from Baseline or Week 1 (depending on when collected) at Week 8 and Week 15
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Attributions of Hostility, Intent, Blame, and Anger (Epps Hypothetical Scenarios) Score
Description: Participants are presented with 21 hypothetical scenarios are 21. After each scenario, participants rate attributions of intent, hostility, and blame, as well as how angry they would be in response to the scenario using a 9-point Likert scale. Scores are calculated for attributions of intent; 2) attributions of hostility; 3) attributions of blame; 4) and anger responses.
  Rating Scale:1,2,3,4,5,6,7,8,9 Scores are calculated for each attribution (intent, hostility, blame) and anger response) Separate average scores are calculated for attributions of intent, hostility, blame and ange.
  Average scores for each range from 1-9. Higher scores indicate more negative attributions or anger.
Time Frame: Change from Baseline at Week 8 and Week 15
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in The Awareness of Social Inference Test (TASIT) Score
Description: The Awareness of Social Inference Test (TASIT) is a performance-based measure that uses short one minute video vignettes to assess emotion recognition and social inferences. Participants' responses are scored as right or wrong. Each correct response earns 1 points. Below are the three subtests that comprise the TASIT. Correct responses are tallied as total scores.
  Part I: Emotion Perception. 28 items. Score ranges from 0-28. Higher score is better performance.
  Part 2: Social inference (minimal context- not much context available to make inference of sincere and sarcastic exchanges). 15 items. Scores range from 0-15. Higher score is better performance.
  Part 3: Social Inference (Enriched context - more context available to make inference of sarcasm and lies). 16 items. Scores range from 0-16. Higher score is better performance.
Time Frame: Change from Baseline at Week 8 and Week 15
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Difficulty With Emotion Regulation Scale (DERS) Score
Description: The Difficulty with Emotion Regulation Scale (DERS) is a 5-point Likert scale that participants use to rate the frequency they utilize self-regulation behaviors in response to general emotional distress.
  Total scores indicate emotion dysregulation or problems with regulating emotions. There are 6 subscales. Subscale scores are summed to generate a total emotion dysregulation score.
  Likert scale (1, 2, 3, 4, 5). Total Raw scores range from 36-180. Higher scores indicate more emotion regulation problems (worse outcome) Subscales are summed to compute a Total Emotion dysregulation raw score.
Time Frame: Change from Week 1 at Week 8 and Week 15
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in The Ambiguous Intentions Hostility Questionnaire (AIHQ) Score
Description: This questionnaire consists of 15 written vignettes describing actions/ situations that were intentional (5), am-biguous (5) and accidental (5). After participants read each vignette and imagine the scenario happening to her or him, they are asked five questions: 1) why the other person (or persons) acted that way toward you (open-ended response later rated by two independent raters; score indicates ''hostility bias''); 2) Whether the other person (or persons) performed the action on purpose (1 ''definitely no'' to 6 ''definitely yes'') using a Likert Scale (Intent score); 3) how angry it would make them feel (1 ''not at all angry'' to 5 ''very angry'') using a Likert scale (anger score); 4) how much they would blame the other person (or persons) (1 ''not at all'' to 5 ''very much'') using a Likert scale (blame score); and 5) how she or he would respond to the situation, (open-ended re-sponse).
Time Frame: Change from Baseline or Week 1(depending on when collected) at Week 8 and Week 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and Serious Adverse events (SAE) were tracked from the time the participant consented to be in the study until their last data collection point (i.e., through study completion). For those randomized to ICAN, this was on average, 4.25 months (range: 2.5 months-8.25 months). For those randomized to WLC, this was on average 6.25 months (range 4.5 months-10.25 months)
Description: ICAN: Because all subjects ultimately received the ICAN intervention (even those who were randomized to WLC), we report AEs and SAEs that occurred surrounding the time of the delivery of ICAN treatment (i.e. during or after treatment delivery) for all 24 enrolled participants.
  WLC: We report AEs and SAEs for those randomized to the WLC arm that occurred prior to treatment delivery (n=14).
Groups:
- WLC: Waitlist Control: WLC participants do not receive treatment until after time two testing 8-weeks from time one testing.
Arm/Group | ICAN | WLC: Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/14
Other Adverse Events (participants affected / at risk) | 12/24 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICAN (N=24) | WLC: Waitlist Control (N=14)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICAN (N=24) | WLC: Waitlist Control (N=14)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject fell and hit head. Went to hospital and had normal MRI results.
scapular dyskinesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin Lupus episode (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) — Both deemed unrelated to study
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 3 (3) | 0 (0)
Flu (Infections and infestations) | 1 (1) | 0 (0)
Perseveration (Psychiatric disorders) | 1 (1) | 0 (0) — Perseveration was probably triggered by study questions.
Bile Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Exhaustion (Social circumstances) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
broken hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Allergies (Infections and infestations) | 0 (0) | 1 (1)
Muscle pain/ body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT03648476/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03648476/ICF_001.pdf